CLINICAL TRIAL: NCT00945477
Title: A Study of Pazopanib as Second Line Therapy in Patients With Metastatic Prostate Cancer Who Have Received Prior Therapy With an LHRH Agonist.
Brief Title: Pazopanib as Second Line Therapy in Patients With Metastatic Prostate Cancer Refractory to Total Androgen Blockade
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Illinois CancerCare, P.C. (Other)
Responsible Party: Principal Investigator, James Knost, Principal Investigator, Illinois CancerCare, P.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILCC #1
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Advanced prostate cancer, treatment, pazopanib (Experimental): Pazopanib
  Interventions: Drug: Pazopanib (GW786034)

INTERVENTIONS:
Drug: Pazopanib (GW786034) — Pazopanib 800 mg daily x 12 weeks
  Other Names: Pazopanib monohydrochloride salt GW786034

SUMMARY:
A growing body of literature supports the role of angiogenesis in the development and spread of a variety of human cancers including prostate cancer.

* Vascular endothelial growth factor (VEGF) expression is low in normal prostate tissue, but markedly increased in tumor tissues, and has a positive association with tumor stage and grade
* Plasma VEGF levels are significantly elevated in patients with hormone refractory prostate cancer (HRPC) compared to those patients with localized disease and have been associated with disease progression in other cancer patient population.
* The Cancer and Leukemic Group-B demonstrated that VEGF levels correlate with survival.

Pazopanib is a potent multi-target receptor tyrosine kinase inhibitor of vascular endothelial growth factor receptors.

DETAILED DESCRIPTION:
VEGF expression is low in all normal prostate tissue, but markedly increased in tumor tissue, and has a positive association with MVD (micro vessel density) tumor stage, grade, and disease-specific survival in patients with prostate cancer. VEGF is known to be under the influence of HIF-1α, which is also up-regulated in the majority of prostate cancer tissue. It has been shown that complete androgen blockade down-regulates VEGF expression via the HIF-1α pathway with concomitant up-regulation of thrombospondin and induction of endothelial cell apoptosis. The VEGF pathway appears to be the dominant vascular formation pathway in prostate cancer with bFGF having a lesser role.

Pazopanib , a hydrochloride salt, is a small molecule inhibitor of several tyrosine kinases, ie: VEGF 1, 2, 3, c-KIT and platelet-derived growth factor receptors. The broad blockade of the VEGF receptors should interfere with the VEGF/VEGF-receptor pathway, and have an impact on cell growth.

According to the NCCN guidelines , first line therapy for metastatic prostate cancer is considered total androgen blockade, either utilizing orchiectomy and/or LH/RH agonists plus Casodex.

Second line therapy would depend on the patient's response to first line therapy, urgency of a response, and the location of metastatic disease.

Pazopanib has been explored in several settings. It has recently been looked at with Bicalutamide in hormone refractory prostate cancer. The second study was with earlier disease, i.e. D-0 relapse androgen-sensitive patients. The University of Chicago has a study looking at the sub-population of prostate cancer patients that have a "chemical relapse" in which patients are given one shot of Lupron, and if the PSA is adequately suppressed, the patients are randomized between pazopanib and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of adenocarcinoma of the prostate histology, currently on total androgen blockage with a bicalutamide.
2. Subjects must provide written informed consent prior to administration of pazopanib or the performance of any study-specific procedures or assessments, and must be willing to comply with treatment and follow up. Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol. Note: It is not necessary that informed consent be obtained within the protocol-specified screening window.
3. Received no prior second line hormone therapy or any chemotherapy. No prior bevacizumab, mTOR inhibitor, sunitinib, sorafenib or other VEGF TKI) for advanced or metastatic prostate cancer.
4. Must have metastatic diagnosis, meaning disease beyond the prostate gland.
5. A progressing PSA of ≥ 3, the PSA will be measured in ≥ 14 days.
6. KPS of ≥ 70
7. Age ≥ 18 years old
8. Adequate organ system functions:

   * Absolute neutrophil count (ANC) ≥ 1.5 X 109/L
   * Hemoglobin ≥ 9 g/dL
   * Platelets ≥ 100 X 109/L
   * International normalized ratio (INR) ≤ 1.2 X upper limit of normal (ULN)
   * Partial thromboplastin time (PTT) ≤ 1.2 X ULN
   * Total bilirubin ≤ 1.5 X ULN
   * AST and ALT ≤ 2.5 X ULN
   * Calculated creatinine clearance ≥ 30 mL/min
   * Urine Protein to Creatinine Ratio (UPC)2 < 1
   * Total serum calcium concentration < 12.0mg/dL

     * Subjects may not have had a transfusion within 7 days of screening assessment.
     * If UPC ≥ 1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value < 1 g to be eligible.
9. Left ventricular ejection fraction (LVEF) ≥ 55% as assessed by echocardiography or multigated acquisition (MUGA) scan. The same modality used at baseline must be applied for subsequent evaluations.

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

1. History of another malignancy.

   Note: Subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
2. History or clinical evidence of central nervous system (CNS) metastases.

   Note: Subjects who have previously-treated CNS metastases (surgery ± radiotherapy, radiosurgery, or gamma knife) and meet all 3 of the following criteria are eligible:
   * Are asymptomatic and,
   * Have had no evidence of active CNS metastases for ≥ 6 months prior to enrollment and,
   * Have no requirement for steroids or enzyme-inducing anticonvulsants (EIAC).
3. Clinically significant gastrointestinal abnormalities including, but not limited to:

   * Malabsorption syndrome,
   * Major resection of the stomach or small bowel that could affect the absorption of study drug,
   * Active peptic ulcer disease,
   * Inflammatory bowel disease,
   * Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation,
   * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
4. Presence of uncontrolled infection.
5. Prolongation of corrected QT interval (QTc) > 480 milliseconds (msecs).
6. History of any one or more of the following cardiovascular conditions within the past 12 months:

   * Cardiac angioplasty or stenting,
   * Myocardial infarction,
   * Unstable angina,
   * Symptomatic peripheral vascular disease,
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA).
7. History of cerebrovascular accident (CVA) including transient ischemic attack (TIA).
8. History of pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anticoagulating agents for at least 6 weeks are eligible.
9. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥150mmHg or diastolic blood pressure (DBP) of ≥ 90 mmHg].

   Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Blood pressure must be re-assessed on two occasions that are separated by a minimum of 24 hours. The mean SBP/DBP values from each blood pressure assessment must be < 150/90mmHg in order for a subject to be eligible for the study. See Section 6.3.2 for instruction on blood pressure measurement and obtaining mean blood pressure values.
10. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
11. Evidence of active bleeding or bleeding diathesis
12. Hemoptysis within 6 weeks of first dose of study drug.
13. Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study.
14. Prohibited medications within 28 days unless the half-life of the medication is longer than 28 days, will not be permitted.
15. Use of an investigational agent, including an investigational anti-cancer agent, within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
16. Prior use of an investigational or licensed drug that targets VEGF or VEGF receptors (e.g., bevacizumab, sunitinib, sorafenib, etc), or are mTOR inhibitors (eg. temsirolimus, everolimus, etc).
17. Is now undergoing and/or has undergone in the last 4 weeks immediately prior to first dose of study drug, (surgery, tumor embolization, chemotherapy, radiation therapy, immunotherapy, or biological therapy)
18. Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity.
19. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Illinois CancerCare, Bloomington, Illinois
  - Illinois CancerCare, Ottawa, Illinois
  - Illinois CancerCare, Pekin, Illinois
  - Illinois Cancer Care, Peoria, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male patients were enrolled from 7/17/2009 through 10/9/2012. All patients were from our practice and screened from our database.
Groups:
- Advanced Prostate Cancer, Treatment, Pazopanib: Pazopanib
  Pazopanib (GW786034) : Pazopanib 800 mg daily x 12 weeks
Period: Overall Study
Arm/Group | Advanced Prostate Cancer, Treatment, Pazopanib
Started | 11
Completed | 5
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Advanced Prostate Cancer, Treatment, Pazopanib
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 68.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Response Rate at 12 Weeks
Description: Response rate defined as 50% decrease in the Prostate Specific Antigen (PSA) level at week 12 compared to baseline
Time Frame: 12 weeks
Population: Five subjects completed the 12 week treatment requirement.
Measure: Number; unit: participants
Groups:
- Pazopanib 800mg Daily by Mouth: Response rate at 12 weeks
Arm/Group | Pazopanib 800mg Daily by Mouth
Number analyzed (Participants) | 5
participants | 2

2. Secondary Outcome: Number Adverse Events, Grades 1-5 Using NCI-CTCAE v 3.0
Description: Safety was evaluated by documentation of Adverse Events (AEs), by assessment of clinical laboratory findings, and by physicial examination, including measurement of vital signs and weight in all eleven subjects.
Time Frame: 0-12 weeks
Population: The adverse events for all participants enrolled were evaluated by documentation of Adverse Events (AEs)Grades 1-5 using NCI-CTCAE v 3.0
Measure: Number; unit: Adverse events Grade 1-5
Groups:
- Participants With Adverse Events 800mg Pazopanib: Adverse events for all participants, all grades
Arm/Group | Participants With Adverse Events 800mg Pazopanib
Number analyzed (Participants) | 11
Adverse events Grade 1-5 | 197

ADVERSE EVENTS:
Time Frame: 0-12 weeks
Arm/Group | Pazopanib 800mg Daily by Mouth
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800mg Daily by Mouth (N=11)
Hemoglobin (Blood and lymphatic system disorders) | 10
Leukocytes (Blood and lymphatic system disorders) | 9
Hypertension (Cardiac disorders) | 8
Fatigue (General disorders) | 10
Anorexia (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 9
Alkaline Phosphatase (Blood and lymphatic system disorders) | 7
AST (SGOT) (Blood and lymphatic system disorders) | 6
Proteinuria (Renal and urinary disorders) | 9
Sodium-serum, low (Blood and lymphatic system disorders) | 7

LIMITATIONS AND CAVEATS:
Because of slow enrollment, the study was terminated. The study planned enrollment of 34 subjects, 11 were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes